CLINICAL TRIAL: NCT02462811
Title: A Double-Blind, Randomized, Active- and Placebo-Controlled, Multiple-Dose, Multi-Center Phase 3 Study of the Safety and Efficacy of CL-108 in the Treatment of Moderate to Severe Pain and Opioid-Induced Nausea and Vomiting (OINV)
Brief Title: A Double-Blind, Randomized, Active- and Placebo-Controlled, Multiple-Dose Multi-Center Phase 3 Study of the Safety and Efficacy of CL-108 in the Treatment of Moderate to Severe Acute Pain and Opioid-Induced Nausea and Vomiting (OINV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Joseph Hazelton (Industry)
Responsible Party: Sponsor-Investigator, Joseph Hazelton, Vice President, Regulatory Affairs, Charleston Laboratories, Inc
Organization: Charleston Laboratories, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCL-003
Record Dates: First submitted 2015-05-22; First posted 2015-06-04 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-01

CONDITIONS: Pain; Nausea; Vomiting
Keywords: Pain; Nausea; Vomiting
MeSH Terms: conditions — Pain; Nausea; Vomiting | interventions — Hydrocodone; Acetaminophen; Promethazine; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CL-108 (Experimental): CL-108 hydrocodone 7.5 mg, acetaminophen 325 mg, Promethazine 12.5 mg
  Interventions: Drug: CL-108 (hydrocodone 7.5 mg, acetaminophen 325 mg, promethazine 12.5 mg)
- Active Comparator: Norco (Active Comparator): Commercial product containing hydrocodone 7.5 mg, acetaminophen 325 mg
  Interventions: Drug: Norco (hyrdocodone 7,5 mg, acetaminophen 325 mg)
- Placebo (Placebo Comparator): CL-108 formulation without API
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CL-108 (hydrocodone 7.5 mg, acetaminophen 325 mg, promethazine 12.5 mg)
  Arms: CL-108
Drug: Placebo
  Arms: Placebo
Drug: Norco (hyrdocodone 7,5 mg, acetaminophen 325 mg)
  Arms: Active Comparator: Norco

SUMMARY:
The objectives of this study are to compare the occurrence and severity of opioid-induced nausea and vomiting (OINV) associated with CL-108 to Norco®, and to demonstrate the efficacy of CL-108 when compared to placebo for the relief of moderate to severe pain In patients with moderate to severe pain following bunionectomy (osteotomy with fixation of the head of the first metatarsal bone).

ELIGIBILITY:
INCLUSION CRITERIA

* Informed Consent: Signed consent obtained at screening prior to any procedures being performed.
* Gender: Male or non-pregnant and non-lactating female. A female of child-bearing potential is eligible to participate in this study if she has a negative urine pregnancy test and is using an acceptable method of birth control (i.e., oral, transdermal, or implanted contraceptives, intrauterine device, diaphragm, condom, abstinence, or surgical sterilization)
* Age: 18 years or older
* OINV Status: At risk of OINV on the Nausea Prone Questionnaire (NPQ)
* Foot Condition: Surgical extraction of a unilateral first metatarsal bunion confirmed by foot x-ray (assessed by surgeon prior to surgery)
* Pain Severity: Presence of moderate or severe pain (i.e., ≥ 4 on the baseline numerical pain intensity rating scale [PI-NRS])
* Pain Confirm: Rating ≥ 50 mm on the baseline visual analog pain intensity scale (PI-VAS)
* Diary Completion: Be willing and able to record safety and efficacy information in the In-patient and Outpatient Diaries
* Safe Transportation: Patient must have arrangements for transportation home from the research center accompanied by a responsible adult

EXLUSION CRITERIA

* Medical Condition: Presence of a serious medical condition (e.g., poorly controlled hypertension or diabetes, neurological disease including Parkinson's or other condition associated with a movement disorder, significantly impaired cardiac, renal, hepatic, respiratory, or thyroid function)
* Infection: Acute local infection at the time of surgery that could confound post-surgical evaluation.
* Drug Allergy: History of hypersensitivity or allergy to an opioid drug such as hydrocodone, promethazine, acetaminophen, ondansetron, NSAID (such as ibuprofen, including aspirin) or ketorolac or history of a dystonic/dyskinetic reaction to prior anti-emetic or anti-psychotic medication
* Contraindicated Drugs: Use (within 24 hours of the surgical procedure) of any confounding prescription or non-prescription drug (e.g., analgesic, anti-emetic, sedating antihistamine, sedative, alcohol, CNS/psychotropic agent, including sleep aides, benzodiazepines, performance/attention enhancers, marijuana, anti-depressants) or any drug contraindicated with hydrocodone, acetaminophen, or promethazine (except for pre-op medications). Antibiotic prophylaxis for endocarditis (except if known to cause nausea) and ASA 62.5 mg for cardiovascular prophylaxis are permitted during the study.
* History of drug or alcohol abuse
* Caffeine Use: Ingestion of any caffeine-containing beverage or chocolate since mid-night before the operation
* Investigation Drug Use: Use of an investigational drug within the past 30 days
* Participated in Study:Previous participation in this study
* Pregnancy, Lactation: Women who are pregnant or lactating
* Participant Relation: Employee at the research center or of Charleston Laboratories or relative of the Principal Investigator, Sub-Investigators, or research staff who is directly involved in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The occurrence of opioid-induced nausea and vomiting (OINV) as assessed by an OINV questionnaire comparing CL-108 to Norco® over 48 hours. | 48 hours
The relief of moderate to severe pain, assessed by visual analog pain intensity scale, comparing CL-108 to placebo over 48 hours (SPID48). | 48 hours

SECONDARY OUTCOMES:
The severity of opioid-induced nausea, comparing CL-108 to Norco® over 48 hours | 48 hours
The occurrence of vomiting, comparing CL-108 to Norco® over 48 hours | 48 hours
The use of anti-emetics, comparing CL-108 to Norco® over 48 hours. | 48 hours
Incidence of post-discharge nausea and vomiting (PDNV), comparing CL-108 to placebo over days 3-5 | 48 hours
The relief of post-operative nausea and vomiting (PONV), comparing CL-108 to placebo over 48 hours | 48 hours
The relief of severe pain, comparing CL-108 to Norco® over 48 hours, i.e., summed pain intensity differences over 48 hours (SPID48) | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Charleston Website — http://www.charlestonlabs.com